CLINICAL TRIAL: NCT02865148
Title: Feasibility and Acceptability of A Behavioral Symptom Management Program for Patients With Advanced Breast Cancer in Singapore and The US
Brief Title: Behavioral Symptom Management Program for Breast Cancer in Singapore and The US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Irene Teo, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DukeNUS
Record Dates: First submitted 2016-07-12; First posted 2016-08-12 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2017-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy (CBT) group (Experimental): Participants will receive 4 sessions that lasts approximately 50 mins. The sessions will teach patients to manage their symptoms.
  Interventions: Behavioral: Cognitive behavioral therapy
- Waitlist control (WLC) group (No Intervention): The WLC group receives standard usual care before being offered the same CBT protocol and assessment thereafter.

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — CBT-based protocol tailored to advanced breast cancer patients with a focus on managing a broad array of symptoms including psychological distress, pain, and fatigue. Important features of the protocol are: 1) a unique motivational interviewing component in the first session that will focus on patients' motivation for engaging in the protocol, confidence (i.e., self-efficacy) to learn new strategies, and potential barriers to adopting recommendations for lifestyle change; and 2) protocol that targets multiple symptoms, and 3) adapted to meet the unique needs of advanced breast cancer patients.
  Arms: Cognitive behavioral therapy (CBT) group

SUMMARY:
Research indicates that up to two-thirds of patients with advanced cancer experience significant symptom burden (e.g., anxiety and depression, pain, fatigue), yet these symptoms are not adequately addressed. Cognitive behavioral therapy (CBT) protocols designed to teach patients strategies to increase their sense of self-efficacy to manage symptoms may be helpful in alleviating multiple cancer-related symptoms. The efficacy of CBT protocols for reducing distinct symptoms in early-stage breast cancer has been shown; however the role of CBT protocols for multiple symptoms in late-stage cancer is less clear. The current study aims to investigate the feasibility and acceptability as well as obtain an initial estimate of efficacy of a novel, cross-cultural CBT intervention that addresses multiple symptoms in advanced breast cancer patients. The target outcomes of intervention will be reduction in symptoms of anxiety and depression, pain, and fatigue. A randomized controlled design will compare patients receiving a CBT protocol to a waitlist control in both Singapore and US patients. The larger goal of this collaborative effort is to determine the scalability of such an intervention that can potentially provide needed symptom burden relief to advanced cancer patients.

DETAILED DESCRIPTION:
Advanced breast cancer refers to metastatic or stage-IV breast cancer, and is associated with the highest cancer mortality and morbidity rates among women. Top symptom complaints reported by patients with advanced breast cancer include fatigue, low mood and worries, and pain. These symptoms frequently co-occur, with presence of stress hormones suggested to be a common mechanism. Greater symptoms of psychological distress (defined as anxiety and depression), pain, and fatigue is associated with decreased quality of life, and adds to the burden and suffering of patients coping with advanced breast cancer. Unfortunately these symptoms are sometimes overlooked and not adequately addressed. This is in turn is associated with increased utilization of healthcare services such as emergency department visits and frequent hospital admissions.

There is a critical need for patients with advanced breast cancer to learn strategies to self-manage common symptoms. Cognitive behavioral therapy (CBT) is a widely used,evidence-based therapy that focuses on cognitions, emotions, and behavior change. The cognitive-behavioral framework has been successfully applied in treatment of many disorders, including anxiety disorders, depression, chronic pain, and insomnia. It is posited that CBT protocols can be designed to meet the needs of advanced breast cancer patients by targeting and modifying maladaptive thoughts about the disease and treatment (e.g., irrational beliefs, unrealistic expectations) and their behavior (e.g., maladaptive coping strategies, isolation, self-negligence). These protocols are designed to teach patients strategies to increase their sense of self-efficacy to manage multiple symptoms may be helpful in alleviating psychological and physical suffering. The efficacy of CBTs for early-stage cancer has been well-documented; however the role of CBTs for late-stage cancer is less clear, particularly in a multi-symptom context. Furthermore, although CBT protocols are more widely used in the US, their use as part of oncologic care in Asia has been limited.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years old
2. Have a diagnosis of stage IV breast cancer
3. Able and willing to attend program sessions
4. Able to speak and read English

Exclusion Criteria:

1. Active serious mental illness (e.g., schizophrenia, bipolar disorder) indicated by medical records
2. Visual, hearing, or cognitive impairment that will interfere with intervention delivery
3. Unaware they have cancer

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Reduction in symptoms of psychological distress | Up to 6 weeks
  Psychological distress will be measured using the Hospital Anxiety Depression Scale (HADS)

SECONDARY OUTCOMES:
Pain level | Up to 6 weeks
  Pain will be measured using the Brief Pain Inventory (BPI)
Fatigue | Up to 6 weeks
  Fatigue will be measured using the PROMIS Fatigue scale

CONTACTS AND LOCATIONS:
Overall Officials: Irene Teo, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Somers TJ, Abernethy AP, Edmond SN, Kelleher SA, Wren AA, Samsa GP, Keefe FJ. A Pilot Study of a Mobile Health Pain Coping Skills Training Protocol for Patients With Persistent Cancer Pain. J Pain Symptom Manage. 2015 Oct;50(4):553-8. doi: 10.1016/j.jpainsymman.2015.04.013. Epub 2015 May 27. PMID 26025279
- [Result] Mahendran R, Lim HA, Tan JY, Chua J, Lim SE, Ang EN, Kua EH. Efficacy of a brief nurse-led pilot psychosocial intervention for newly diagnosed Asian cancer patients. Support Care Cancer. 2015 Aug;23(8):2203-6. doi: 10.1007/s00520-015-2771-0. Epub 2015 May 23. PMID 26001988